CLINICAL TRIAL: NCT05502341
Title: An Operationally Seamless Phase 2/3 Randomized, Open-label, Multicenter, Active-Controlled Study to Evaluate the Safety and Efficacy of Bictegravir/Lenacapavir Versus Stable Baseline Regimen in Virologically Suppressed People With HIV-1 on Stable Complex Treatment Regimens
Brief Title: Study to Compare Bictegravir/Lenacapavir Versus Current Therapy in People With HIV-1 Who Are Successfully Treated With a Complicated Regimen
Acronym: ARTISTRY-1
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-621-6289; 2022-500929-33 (Other: European Medicines Agency); DOH-27-052023-8574 (Other: South African Clinical Trial Registry); jRCT2051230168 (Other: Japan registry)
Record Dates: First submitted 2022-08-05; First posted 2022-08-16 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — bictegravir; lenacapavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 2: Bictegravir (BIC) 75 mg + Lenacapavir (LEN) 25 mg (Experimental): Participants will switch from their stable baseline regimen (SBR) to a regimen of BIC 75 mg + LEN 25 mg. Participants will receive a 2-day loading dose regimen of LEN 600 mg, in addition to the daily doses of BIC 75 mg + LEN 25 mg starting on Day 1 up to the end of randomized treatment (ERT) visit, participants will be treated for at least 24 weeks during the Randomized Period.
  Following Randomized Period, the participants will have an option to participate in an Extension Period to receive BIC/LEN 75 mg/50 mg fixed dose combination (FDC).
  Interventions: Drug: Bictegravir; Drug: Lenacapavir
- Phase 2: BIC 75 mg + LEN 50 mg (Experimental): Participants will switch from their SBR to a regimen of BIC 75 mg + LEN 50 mg. Participants will receive a 2-day loading dose regimen of LEN 600 mg, in addition to the daily doses of BIC 75 mg + LEN 50 mg starting on Day 1 up to the ERT visit, participants will be treated for at least 24 weeks during the Randomized Period.
  Following Randomized Period, the participants will have an option to participate in an Extension Period to receive BIC/LEN 75 mg/50 mg FDC.
  Interventions: Drug: Bictegravir; Drug: Lenacapavir
- Phase 2: Stable Baseline Regimen (SBR) (Active Comparator): Participants will continue with their SBR per prescription for up to the ERT visit, participants will be treated for at least 24 weeks during the Randomized Period.
  Following Randomized Period, the participants will have an option to participate in an Extension Period to receive BIC/LEN 75 mg/50 mg FDC.
  Interventions: Drug: Stable Baseline Regimen
- Phase 3: BIC/LEN 75 mg/50 mg Fixed-dose Combination (FDC) (Experimental): Participants will switch from their SBR to a regimen of BIC/LEN 75 mg/50 mg FDC. Participants will receive a 2-day loading dose regimen of LEN 600 mg, in addition to the daily doses of BIC/LEN 75 mg/50 mg FDC starting on Day 1 up to the ERT visit, participants will be treated for at least 48 weeks during the Randomized Period.
  Following Randomized Period, the participants will have an option to participate in an Extension Period to receive BIC/LEN 75 mg/50 mg FDC.
  Interventions: Drug: BIC/LEN FDC
- Phase 3: Stable Baseline Regimen (Active Comparator): Participants will continue with their SBR per prescription for up to the ERT visit, participants will be treated for at least 48 weeks during the Randomized Period.
  Following Randomized Period, the participants will have an option to participate in an Extension Period to receive BIC/LEN 75 mg/50 mg FDC.
  Interventions: Drug: Stable Baseline Regimen

INTERVENTIONS:
Drug: Bictegravir — Tablets administered orally without regard to food
  Other Names: GS-9883
  Arms: Phase 2: BIC 75 mg + LEN 50 mg; Phase 2: Bictegravir (BIC) 75 mg + Lenacapavir (LEN) 25 mg
Drug: Lenacapavir — Tablets administered orally without regard to food
  Other Names: GS-6207
  Arms: Phase 2: BIC 75 mg + LEN 50 mg; Phase 2: Bictegravir (BIC) 75 mg + Lenacapavir (LEN) 25 mg
Drug: BIC/LEN FDC — Tablets administered orally without regard to food
  Arms: Phase 3: BIC/LEN 75 mg/50 mg Fixed-dose Combination (FDC)
Drug: Stable Baseline Regimen — SBR will include a combination of antiretroviral (ARV) regimen. ARV regimen may include the following, except for participants taking a single tablet regimen or taking a complete parenteral regimen (Cabenuva).
  * Nucleos(t)ide Reverse Transcriptase Inhibitors:
    * Abacavir
    * Emtricitabine
    * Lamivudine
    * Tenofovir alafenamide
    * Tenofovir disoproxil fumarate
    * Zidovudine
  * Non-Nucleosite Reverse Transcriptase Inhibitors:
    * Delavirdine
    * Efavirenz
    * Nevirapine
    * Rilpivirine
    * Doravirine
  * Integrase Inhibitors:
    * Bictegravir
    * Cabotegravir
    * Dolutegravir
    * Elvitegravir
    * Raltegravir
  * Protease Inhibitors:
    * Atazanavir
    * Darunavir
    * Fosamprenavir
    * Indinavir
    * Lopinavir
    * Nelfinavir
    * Saquinavir
    * Tipranavir
  * Chemokine Co-receptor 5 (CCR5) Antagonist:
    * Maraviroc
  * Fusion Inhibitors:
    * Enfuvirtide
  * gp120 Attachment Inhibitor:
    * Fostemsavir
  * Anti-CD4 Monoclonal Antibodies:
    * Ibalizumab-uiyk
  Arms: Phase 2: Stable Baseline Regimen (SBR); Phase 3: Stable Baseline Regimen

SUMMARY:
The goal of this clinical study is to learn more about the effects of switching to the study drugs, bictegravir (BIC) plus lenacapavir (LEN), versus current therapy (Phase 2) and BIC/LEN fixed-dose combination (FDC) versus current therapy (Phase 3) in people living with HIV (PWH).

ELIGIBILITY:
Key Inclusion Criteria:

* If plasma HIV-1 RNA measurements in the 6 months prior to screening are available, all levels must be < 50 copies/mL.
* At least one documented plasma HIV-1 RNA level measured between 6 and 12 months (± 2 months) prior to screening. This and any other HIV-1 RNA measurements documented in this period must be < 50 copies/mL
* Plasma HIV-1 RNA levels < 50 copies/mL at screening.
* Currently receiving a complex antiretroviral (ARV) regimen due to previous viral resistance, or intolerance, or contraindication to existing single-tablet regimens (STR), and on this regimen for at least 6 months prior to the screening visit. The criteria to define a complex regimen in this study are as follows:

  * A regimen containing a boosted protease inhibitor or a nonnucleos(t)ide reverse transcriptase inhibitor (NRTI) plus at least 1 other third agent (ie, an agent from a class other than NRTIs) (eg, bictegravir/emtricitabine/tenofovir alafenamide (coformulated; Biktarvy®)(BVY) + darunavir/cobicistat, BVY + etravirine), or
  * A regimen of ≥ 2 pills/day, or a regimen requiring dosing more than once daily, or
  * A regimen containing parenteral agent(s) (excluding a complete long-acting injectable regimen, such as intramuscular cabotegravir plus rilpivirine) as well as oral agents.
* No documented or suspected resistance to bictegravir (BIC).
* Estimated glomerular filtration rate ≥ 15 mL/min according to the Cockcroft-Gault formula for creatinine clearance (CLcr) who are not on renal replacement therapy.

Key Exclusion Criteria:

* Prior use of, or exposure to, lenacapavir (LEN)
* Active tuberculosis infection
* Chronic hepatitis B virus (HBV) infection

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 689 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Phase 2: Proportion of Participants With HIV-1 RNA ≥ 50 Copies/mL at Week 24 as Determined by the US FDA-defined Snapshot Algorithm | Week 24
Phase 3: Proportion of Participants With HIV-1 RNA ≥ 50 Copies/mL at Week 48 as Determined by the US FDA-defined Snapshot Algorithm | Week 48

SECONDARY OUTCOMES:
Phase 2: Proportion of Participants With HIV-1 RNA < 50 Copies/mL at Week 24 as Determined by the US FDA-defined Snapshot Algorithm | Week 24
Phase 2: Change From Baseline in CD4 Cell Count at Week 24 | Baseline, Week 24
Phase 2: Percentage of Participants Experiencing Treatment-emergent Adverse Events (AEs) Through Week 24 | First dose date up to Week 24
Phase 2: Pharmacokinetic (PK) Parameter: Cmax of Bictegravir (BIC) and Lenacapavir (LEN) at Steady State | Day 1 up to Week 24
  Cmax is defined as the maximum observed concentration of drug.
Phase 2: PK Parameter: AUCtau of BIC and LEN at Steady State | Day 1 up to Week 24
  AUCtau is defined as the area under the concentration versus time curve over the dosing interval.
Phase 2: PK Parameter: Ctau of BIC and LEN at Steady State | Day 1 up to Week 24
  Ctau is defined as the observed drug concentration at the end of the dosing interval.
Phase 3: Proportion of Participants With HIV-1 RNA < 50 Copies/mL at Week 48 as Determined by the US FDA-defined Snapshot Algorithm | Week 48
Phase 3: Change From Baseline in CD4 Cell Count at Week 48 | Baseline, Week 48
Phase 3 (BIC/LEN 75 mg/50 mg FDC): Proportion of Participants from With HIV-1 RNA ≥ 50 Copies/mL at Week 96 as Determined by the US FDA-defined Snapshot Algorithm | Week 96
Phase 3 (BIC/LEN 75 mg/50 mg FDC): Change From Baseline in CD4 Cell Count at Week 96 | Baseline, Week 96
Phase 3: Percentage of Participants Experiencing Treatment-emergent AEs Through Week 48 | First dose date up to Week 48
Phase 3 (BIC/LEN 75 mg/50 mg FDC): Proportion of Participants from Experiencing Treatment-emergent AEs Through Week 96 | Week 96

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (93):
- United States (40):
  - Be Well Medical Center, Berkeley, California
  - Pacific Oaks Medical Group, Beverly Hills, California
  - Ruane Clinical Research Group, Inc, Los Angeles, California
  - Alta Bates Summit Medical Center, Summit Campus, East Bay Advanced Care, Oakland, California
  - Bios Clinical Research, Palm Springs, California
  - University of California San Diego (UCSD), San Diego, California
  - Lundquist Institute for Biomedical Innovation at Harbor - UCLA Medical Center, Torrance, California
  - The Men's Health Foundation, West Hollywood, California
  - Denver Health Medical Center, Denver, Colorado
  - Yale University; School of Medicine; AIDS Program, New Haven, Connecticut
  - Midland Florida Clinical Research Center, LLC, DeLand, Florida
  - Therafirst Medical Centers, Fort Lauderdale, Florida
  - Gary Richmond, MD, PA, Inc., Fort Lauderdale, Florida
  - Midway Immunology & Research Center, LLC, Ft. Pierce, Florida
  - Schiff Center for liver Diseases/University of Miami, Miami, Florida
  - Floridian Clinical Research, Miami Lakes, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Therapeutic Concepts, PA, Orlando, Florida
  - Triple O Research Institute PA, West Palm Beach, Florida
  - Atlanta ID Group, Atlanta, Georgia
  - Mercer University School of Medicine, Macon, Georgia
  - Howard Brown Health Center, Chicago, Illinois
  - Kansas City Care Clinic, Kansas City, Missouri
  - Southampton Healthcare, Inc., St Louis, Missouri
  - Saint Michael's Medical Center, Newark, New Jersey
  - AXCES Research Group, Santa Fe, New Mexico
  - New York Presbyterian Hospital, Flushing, New York
  - Ricky K. Hsu, MD, PC, New York, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Medical University of South Carolina (MUSC) Research NEXUS, Charleston, South Carolina
  - Central Texas Clinical Research, Austin, Texas
  - St. Hope Foundation, Bellaire, Texas
  - AIDS Arms, Inc., DBA Prism Health North Texas, Dallas, Texas
  - North Texas Infectious Diseases Consultants, Dallas, Texas
  - Texas Centers for Infectious Disease Associates, Fort Worth, Texas
  - Gordon E. Crofoot MD PA, Houston, Texas
  - Diagnostic Clinic of Longview - Center for Clinical Research, Longview, Texas
  - Peter Shalit, MD, Seattle, Washington
- Argentina (3):
  - Hospital General de Agudos J.M Ramon Mejia, Buenos Aires
  - Fundación Huésped, Buenos Aires
  - Helios Salud, Buenos Aires
- Australia (4):
  - St.Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Taylor Square Private Clinic, Darlinghurst, New South Wales
  - Holdsworth House Medical Practice, Sydney, New South Wales
  - Alfred Health, Melbourne, Victoria
- Canada (6):
  - Chronic Viral Illness Service / McGill University Health Centre (MUHC), Decarie Montreal
  - Clinique Medicale du Quartier Latin, Montreal
  - The Ottawa Hospital - General Campus, Ottawa
  - ID Clinic, Regina
  - Maple Leaf Research, Toronto
  - Spectrum Health, Vancouver
- Instituto Dominicano de Estudio Virologicos - IDEV, Santo Domingo, Dominican Republic
- France (4):
  - CHU Nice-Hôpital l'Archet, Nice
  - Hospital Saint Louis, Paris
  - Groupe Hospitalier Bichat Claude Bernard, Paris
  - Höpital de la Pitié Salpêtrière, Paris
- Germany (5):
  - zibp Zentrum für Infektiologie Berlin Prenzlauer Berg GmbH, Berlin
  - Universitatsklinikum Bonn, Bonn
  - Infektio Research GmbH & Co.KG, Frankfurt
  - ICH Study Center GmbH & Co. KG, Hamburg
  - MVZ München am Goetheplatz, München
- Italy (5):
  - IRCCS Ospedale San Raffaele, Milan
  - ASST Fatebenefratelli Sacco, Milan
  - Azienda Ospedaliero-Universitaria di Modena, Modena
  - Istituto Nazionale Malattie Infettive "Lazzaro Spallanzani" IRCCS, Roma
  - ASL Città di Torino, Torino
- Japan (3):
  - National Hospital Organization Nagoya Medical Center, Nagoya
  - National Hospital Organization Osaka National Hospital, Osaka
  - Center Hospital of the National Center for Global Health and Medicine, Tokyo
- Puerto Rico (2):
  - Hope Clinical Research, San Juan, PR
  - Proyecto ACTU, San Juan, PR
- South Africa (3):
  - Desmond Tutu Health Foundation Clinical Trials Unit, Cape Town
  - Sefako Makgatho Health Sciences University, Ga-Rankuwa
  - Ezintsha, Johannesburg
- South Korea (4):
  - Kyungpook National University Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Yonsei University Severance Hospital, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
- Spain (5):
  - Hospital Clinic Provincial de Barcelona, Barcelona
  - Hospital Ramon y Cajal, Madrid, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
- Taiwan (3):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - Taoyuan General Hospital, Taoyuan
- United Kingdom (5):
  - Department of HIV & Sexual Medicine, Birmingham
  - Brighton and Sussex University Hospitals NHS Trust, Brighton
  - Barts Health NHS Trust, London
  - HIV medicine and infectious diseases, London
  - St.Stephen's AIDS Trust, Clinical Trials Unit, 1st Floor, St.Stephen's Centre, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-621-6289